CLINICAL TRIAL: NCT06623383
Title: Correlation of Fecal Calprotectin and Fecal Immunochemical Test in Determination of Endoscopic Activity in Inflammatory Bowel Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Associate professor, Mahidol University
Other Study IDs: 579/2566(IRB2)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; inflammatory bowel disease; endoscopy; fecal calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease (IBD) patients often experience a long disease course with periods of remission and flare-ups. Currently, in addition to assessing disease stages based on symptoms, colonoscopy performed by specialized physicians is considered the standard for accurately monitoring disease activity. This procedure allows direct visualization of intestinal lesions. However, colonoscopy is complex, costly, carries the risk of complications, and is not suitable for frequent monitoring. This study aims to explore whether stool tests such as calprotectin and immunochemical tests, which are now standard for assessing disease activity in IBD, correlate with colonoscopy results. It also aims to assess the efficacy of these stool tests in determining whether the disease is in remission or active.

The objective of the study is to investigate the correlation and efficacy of stool test results, calprotectin and fecal immunochemical test, compared to colonoscopy in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Diagnosed with inflammatory bowel disease, either ulcerative colitis or Crohn's disease.
* Scheduled for colonoscopy for various indications, including:

  1. Follow-up after treatment to assess disease remission
  2. Clinical symptoms or laboratory results suggesting disease flare, such as increased abdominal pain, more frequent diarrhea, or elevated inflammatory markers in the blood
  3. Screening for colorectal cancer in patients with long-standing inflammatory bowel disease.

Exclusion Criteria:

* Patients who decline participation in the research project. Incomplete or unsuccessful colonoscopy.
* Failure to provide stool samples.
* Patients hospitalized for reasons unrelated to inflammatory bowel disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients follow-up at Siriraj Hospital, Bangkok, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To study the correlation between fecal calprotectin and fecal immunochemical test for hemoglobin results and endoscopic scores from colonoscopy in patients with inflammatory bowel disease | 1 year
  To study the correlation between fecal calprotectin and fecal immunochemical test for hemoglobin results and endoscopic scores from colonoscopy in patients with inflammatory bowel disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No